CLINICAL TRIAL: NCT05698537
Title: Risk Factors and Etiologies of Epilepsy in Urban and Rural Rwanda
Acronym: REpiCa
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2022-0403
Record Dates: First submitted 2023-01-04; First posted 2023-01-26 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Epilepsy
Keywords: Epilepsy; Epilepsy / etiology; Epilepsy / epidemiology; Seizures; Africa South of the Sahara; Risk Factors; Case-Control Studies
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Electroencephalography; Neuroimaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People living with epilepsy (PwE): Study participants with epilepsy
  Interventions: Diagnostic Test: EEG; Diagnostic Test: Neuroimaging; Diagnostic Test: Blood sample; Other: Risk factor questionnaire
- Control subjects: Study participants without epilepsy
  Interventions: Diagnostic Test: Blood sample; Other: Risk factor questionnaire

INTERVENTIONS:
Diagnostic Test: EEG — EEG registration performed in PwE to confirm epilepsy diagnosis
  Groups: People living with epilepsy (PwE)
Diagnostic Test: Neuroimaging — Neuroimaging performed in PwE to diagnose epilepsy etiology
  Other Names: CT/MRI
  Groups: People living with epilepsy (PwE)
Diagnostic Test: Blood sample — Blood samples from both PwE and controls will be collected to measure full blood count, IgM and IgG antibodies to parasitic antigens including Taenia solium, Toxoplasma gondii and Plasmodium falciparum, to perform ELISA for HIV1 and HIV2, to measure HIV viral load and to conduct an emmel test.
Other: Risk factor questionnaire — Both PwE and control subjects will complete a structured questionnaire on a wide range of potential risk factors present before the onset of the epilepsy.

SUMMARY:
Epilepsy is one of the most common chronic brain disorders. Up to 85% of persons living with epilepsy (PwE) live in the developing world. In sub-Saharan Africa (SSA), Rwanda has one of the highest prevalence rates (±5%). Higher prevalence in low-and middle-income countries (LMICs) can partly be attributed to differences in risk factors for epilepsy of which a great number are preventable. Expanding knowledge on risk factors and etiologies of epilepsy in Rwanda can lower the portion of preventable epilepsies and decrease the high number of Rwandan PwE. This project will focus on the investigation of risk factors and etiologies of epilepsy in urban and rural Rwanda using a nationwide approach.

DETAILED DESCRIPTION:
Risk factors and etiologies of epilepsy in the Rwandan population will be determined using two phases. The initial phase (Task 1) includes the recruitment of the study population using two separate surveys. The first survey (Task 1.1.) will be conducted in the general population by a door-to-door (D2D) approach. During D2D visits in 10 selected urban and rural villages throughout the country, one rural and one urban per province, persons of the households with permanent residence will be interviewed by enumerators to screen for epilepsy. In case of a positive screening, they will be assessed by a team of Rwandan and Belgian neurologists to confirm the epilepsy diagnosis. During a second survey (Task 1.2.), PwE will be matched with control persons defined as persons who screened negative during the Task 1.1 survey.

The second phase of our study (Task 2) consists of the assessment of potential risk factors associated with epilepsy using the matched case-control group (Task 2.1.), and the identification of underlying etiology in PwE according to the International League Against Epilepsy (ILAE) etiology guidelines (Task 2.2.).

Task 2.1. Both cases and controls will complete a structured questionnaire on a wide range of potential risk factors present before the onset of the epilepsy, administered by research assistants. In addition, blood samples from both PwE and controls will be collected as to measure the exposure to parasitic infections and HIV, and the presence of sickle cell disease, among others. Exposure will be measured by detection of IgG antibodies to parasitic antigens including Taenia solium, Toxoplasma gondii and Plasmodium falciparum as well as HIV in plasma samples of the participants.

Task 2.2. Further, in order to classify PwE according to the ILAE etiology guidelines, we will use the detailed medical and epilepsy history including in-depth narrative of seizure description and frequency, clinical examination and narrative of epilepsy treatment assessed by the team of neurologists subsequent to the confirmation of the epilepsy diagnosis. In addition, all PwE will undergo EEG recording using a mobile device. Furthermore, PwE will undergo CT- or MRI-imaging unless previous imaging studies have been performed and are accessible for re-evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Inhabitants of the selected villages who screen positive on the Limoges epilepsy screening questionnaire during the D2D visits and have a confirmed epilepsy diagnosis assessed by a team of Rwandan and Belgian neurologists, are included as PwE. Epilepsy will be defined as unprovoked recurrent seizures occurring more than 24h apart, including active and lifetime epilepsy.
* Persons with a negative screening during the D2D visits who match with a PwE for age and gender and have an absence of epilepsy confirmed during a clinical assessment by a team of Rwandan and Belgian neurologists, are included as control persons.

Exclusion Criteria:

* Inhabitants of the selected villages who are unwilling to complete a verbal witnessed informed consent during D2D visits. For patients ≤18 years of age, verbal consent will be obtained from their parents/caregivers.
* PwE and selected control persons who are unwilling to sign a written informed consent upon referral for neurological assessment.
* PwE and control persons not meeting the inclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be recruited using two surveys. The first survey (Task 1.1.) will be conducted in the general population of the 10 selected villages. Persons of the households with permanent residence will be interviewed by enumerators during door-to-door visits using the Limoges epilepsy screening questionnaire. If a person screens positive, they will be assessed by a team of Rwandan and Belgian neurologists to confirm epilepsy diagnosis. Subsequently, PwE will be matched with control persons through a second survey (Task 1.2.). Persons with a negative screening during the first survey who match for age and gender will be contacted for a clinical assessment by Rwandan and Belgian neurologists to confirm absence of epilepsy. Final matching will have a ratio 1:1.
Sampling Method: Probability Sample
Enrollment: 1745 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Association between epilepsy and exposure of possible risk factors for epilepsy | Baseline
  The following risk factors will be assessed in both PwE and control subjects: family history of seizures, history of febrile seizures, history of head trauma, history of CNS infections and tuberculosis, history of perinatal events, cassava consumption and malnutrition, immunization status against common communicable diseases, history of cerebrovascular disease including hypertension, hypercholesterolemia and diabetes mellitus as primary risk factors and consumption of alcohol, drugs and tobacco; using a risk factor questionnaire. Additional risk factors including exposure to parasitic infections e.g., toxoplasmosis, malaria, neurocysticercosis and HIV, and the presence of sickle cell disease, among others, will be measured by analysis of blood samples. Primary risk factors associated with the mentioned parasitic infections and HIV are included in the questionnaire.
Etiologies of epilepsy | Baseline
  Etiologies of epilepsy in PwE will be classified according to the 2017 International League Against Epilepsy (ILAE) criteria using detailed medical and epilepsy history, clinical examination and paraclinical investigations including EEG recording and neuroimaging in PwE only.

SECONDARY OUTCOMES:
Male and female epilepsy risk factors and etiologies | Baseline
  A sub-analysis comparing male and female epilepsy risk factors and etiologies will be conducted.
Prevalence of epilepsy | Baseline
  Establishment of prevalence of epilepsy in selected villages
Diagnosis gap | Baseline
  Previous diagnosis of epilepsy if applicable, including who initially made the diagnosis and when, will be self-reported during epilepsy screening in the selected villages defining newly and previously diagnosed patients (diagnosis gap).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, MD-PhD, Study Chair — University Hospital, Ghent; Dirk Teuwen, MD, Study Director — University Hospital, Ghent; Ieme Garrez, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- King Faisal Hospital, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Anonymized, analytical datasets and statistical outputs as well as final study documents including figures and tables will be offered for deposit to 4TU.ResearchData, which is a certified data repository accepting research data in the field of medicine and health care and preserving them for a minimum of 15 years.
Time Frame: Data will be made available upon publication of the research results.
Access Criteria: Open Access repository
URL: https://data.4tu.nl/info/en/

REFERENCES:
- [Background] Dedeken P, Sebera F, Mutungirehe S, Garrez I, Umwiringirwa J, Van Steenkiste F, Boon PAJM, Teuwen DE. High prevalence of epilepsy in Northern Rwanda: Exploring gender differences. Brain Behav. 2021 Nov;11(11):e2377. doi: 10.1002/brb3.2377. Epub 2021 Oct 17. PMID 34661989
- [Background] Sebera F, Munyandamutsa N, Teuwen DE, Ndiaye IP, Diop AG, Tofighy A, Boon P, Dedeken P. Addressing the treatment gap and societal impact of epilepsy in Rwanda--Results of a survey conducted in 2005 and subsequent actions. Epilepsy Behav. 2015 May;46:126-32. doi: 10.1016/j.yebeh.2015.03.028. Epub 2015 Apr 30. PMID 25936276